CLINICAL TRIAL: NCT01095107
Title: Relationship of Energy Density of Foods Within a Nutritional Insufficiency Patient's Diet to Inpatient Hospital Stay Duration, Body Image, Mood and Gastrointestinal Symptoms
Brief Title: Food Energy Density in Eating Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Couldn't offer patients a high/low fat meal plan because food service changes
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ellen Rome, Staff, General Pediatrics, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CCCH-KW
Record Dates: First submitted 2010-03-19; First posted 2010-03-29 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Nutritional Insufficiency
Keywords: Determining whether adjustments in the amounts of fat grams within the current inpatient protocol meal plans will lead to a change in the hospital stay duration; Alter their recovery by affecting vital signs; Rate of weight change or need for supplemental feeds/medications; Effect gastrointestinal symptoms (bloating, gastroesophageal reflux, constipation, diarrhea, abdominal pain; And/or effect their perceived body image or cause any changes in their mood.
MeSH Terms: conditions — Gastroesophageal Reflux; Constipation; Diarrhea; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm = Decreased Energy Density (Other): Decreased energy density = 35-50 grams of fat per day between meals and snacks
  Interventions: Dietary Supplement: Low fat intake
- Treatment Arm = Increased Energy Density (Other): increased increased energy density : Intake > 50 grams of fat per day between meals and snacks
  Interventions: Dietary Supplement: Increased fat intake

INTERVENTIONS:
Dietary Supplement: Low fat intake — low fat intake : Intake 35-50 grams of fat per day between meals and snacks
  Arms: Control Arm = Decreased Energy Density
Dietary Supplement: Increased fat intake — increased fat intake : Intake > 50 grams of fat per day between meals and snacks
  Arms: Treatment Arm = Increased Energy Density

SUMMARY:
Nutritional insufficiency is defined as an inadequate amount of nutrition due to decreased food/caloric intake, often due to an eating disorder, such as anorexia nervosa or bulimia. Often when re-feeding these chronically malnourished patients, they can experience changes in their mood and/or body image, metabolic abnormalities and functional aberrations of their gastrointestinal system described as re-feeding syndrome, which all can adversely effect their recovery. In our pilot study, we are attempting to determine whether adjustments in the amounts of energy dense foods, such as fat, in the current inpatient protocol meal plans will lead to a change in the hospital stay duration, alter their recovery by affecting vital signs, weight or need for supplemental feeds or medications, effect gastrointestinal re-feeding syndrome symptoms (bloating, gastroesophageal reflux, constipation, diarrhea, abdominal pain), and/or effect their perceived body image or cause any changes in their mood.

1. To determine whether a higher amount of fat calories per day within a normal range in a Nutritional Insufficiency patient's diet will lead to a shorter inpatient hospital stay duration.
2. To determine whether a higher amount of fat calories per day within a normal range in a Nutritional Insufficiency patient's diet will lead to less gastrointestinal re-feeding syndrome symptoms.
3. To determine whether a higher amount of fat calories per day within a normal range in a Nutritional Insufficiency patient's diet will effect their body image and/or alter their mood.

DETAILED DESCRIPTION:
A randomized, double blind pilot study; physicians and patients will be blinded as to which treatment group they will be placed, nutrition therapists will perform randomization and placement into each treatment group for this research study, along with the development of daily meal plan as they typically do when not involved in this study, and therefore they will not be blinded.

Research Procedures

Patients will be placed into one of two groups:

1. Control: Intake 35-50 grams of fat per day between meals and snacks - this is the typical amount used within our current inpatient re-feeding meal plan, still within a healthy range as it is at the lower end of normal, which given that these patients typically consume a "low fat" diet prior to admission that this amount has been the standard of care for treatment thus far, if they require any supplemental feedings for incomplete meals it will be with the standard lower fat content supplements
2. Treatment: Intake > 50 grams of fat per day between meals and snacks - still within a healthy range as it is at the higher end of normal, if they require any supplemental feedings for incomplete meals it will be with a higher fat content supplement as dictated by the nutrition therapists

Study instruments - questionnaires distributed and collected on the initial day of admission, on every third day of inpatient stay and on the day of discharge by the nutrition therapists. Due to the lack of research on this method of treatment, there are no questionnaires which have been tested for validity and reliability; therefore we have created our own, which we plan to assess during this pilot study. We also plan to follow-up with the patient and parent(s) at 1 month post-discharge (+/- 1 day) to assess how their re-feeding treatment has been going, along with to assess how they feel and ask about any symptoms they are experiencing.

Tests and procedures - all patients with Nutritional Insufficiency/Eating Disorders admitted to the Cleveland Clinic Children's Hospital follow the Nutritional Insufficiency Protocol, with all screening tests and inpatient evaluation and follow-up occurring regardless of whether they are involved in the current pilot study. As per protocol, these patients will be on strict bed rest with a 24 hour companion supervising the patient at all times, especially monitoring intake and timing of completion of all meals, snacks and/or supplements. It is also standard per protocol that they receive Neutra-phos which is a potassium phosphate and sodium phosphate supplement, twice daily for the initial 5 days of treatment. The screening, daily inpatient evaluation, and study questionnaire distribution will be completed on admission, every 3 days, and at discharge

ELIGIBILITY:
Inclusion Criteria:

• Males and females < 25 years of age admitted through the Adolescent Medicine service for inpatient treatment of Nutritional Insufficiency/Eating Disorder or any significant medical abnormalities associated with Nutritional Insufficiency/Eating Disorder.

Exclusion Criteria:

* Elevated liver function tests,
* Elevated pancreatic enzymes,
* Expected admission < 24 hours duration,
* Admission on weekends.

Ages: 9 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 1 year
Blood pressure | 1 year
Weight Changes | 1 year
Need for constipation medications | 1 year
Need for supplemental nutrition | 1 year
Need for reflux medications | 1 year
Bloating Symptoms | 1 year
Constipation symptoms | 1 year
Gastroesophageal reflux symptoms | 1 year
Perceived body image | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Rome, MD, Principal Investigator — The Cleveland Clinic